CLINICAL TRIAL: NCT03305159
Title: Tolerance of Chlorhexidine Gluconate Versus Povidone Iodine Vaginal Cleansing Solution: a Randomized Control Trial
Brief Title: Tolerance of Chlorhexidine Gluconate Vaginal Cleansing Solution
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Magdy Milad, MD, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STU00204759
Record Dates: First submitted 2017-09-04; First posted 2017-10-09 (Actual); Results first posted 2019-06-27 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Surgical Preparation of the Vagina
MeSH Terms: interventions — Povidone-Iodine; chlorhexidine gluconate

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomized to either the control (povidone iodine) or intervention (chlorhexidine gluconate).
Who Masked: Participant
Masking Description: Patients will be randomized to the control or intervention and not be told which antiseptic they received for the surgical preparation of the vagina.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (Povidone Iodine) (Active Comparator): Patients to receive povidone iodine for the surgical preparation of the vagina.
  Interventions: Drug: Povidone-Iodine
- Intervention (4% Chlorhexidine gluconate) (Experimental): Patients to receive 4% chlorhexidine gluconate for the surgical preparation of the vagina.
  Interventions: Drug: 4% Chlorhexidine Gluconate

INTERVENTIONS:
Drug: Povidone-Iodine — Patients will receive povidone iodine for the surgical preparation of the vagina.
  Arms: Control (Povidone Iodine)
Drug: 4% Chlorhexidine Gluconate — Patients will receive 4% chlorhexidine gluconate for the surgical preparation of the vagina.
  Arms: Intervention (4% Chlorhexidine gluconate)

SUMMARY:
Conduct a randomized control study to compare the tolerance of 4% chlorhexidine gluconate/4% isopropyl alcohol versus povidone iodine vaginal cleansing solutions for surgical preparations of the vagina. Patients will be randomized to either control (povidone iodine) or experimental (chlorhexidine gluconate), and then be given a short survey prior to and immediately after surgery, and again 24-48 hours via phone asking them about the presence and severity of vaginal dryness, burning, itchiness, unusual vaginal discharge, and pain or burning with urination.

DETAILED DESCRIPTION:
Surgical site antisepsis is critical in preventing surgical site infections. Although chlorhexidine gluconate has proven to be superior to povidone iodine for surgical site antisepsis, povidone iodine is the only FDA-approved antiseptic solution for surgical preparation of the vagina. Many surgeons are hesitant to use chlorhexidine gluconate for preoperative vaginal cleansing due to the alcohol dissolvent present in the solutions that is implicated in a greater risk of irritation. Yet, there has been no randomized study to illustrate whether the risk of vaginal irritation is greater in chlorhexidine gluconate versus povidone iodine. Thus, the purpose of the study is to conduct a randomized control trial to compare the tolerance of 4% chlorhexidine gluconate to povidone iodine using patient-reported outcomes of vaginal or urinary symptoms. Patients will be randomized to either control or experimental, and then be given a short survey prior to and immediately after surgery, and again 24-48 hours via phone asking them about the presence and severity of vaginal dryness, burning, itchiness, unusual vaginal discharge, and pain or burning with urination.

ELIGIBILITY:
Inclusion Criteria:

1. Undergoing hysteroscopy
2. Gynecologic dilation & curettage
3. Endometrial ablation
4. Essure without concomitant laparoscopy

Exclusion Criteria:

1. Pregnant
2. Have a history of atopic dermatitis, vaginal irritation, allergic reactions, or anaphylaxis to chlorhexidine gluconate or povidone iodine.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Magdy Milad, MD, Principal Investigator — Northwestern University
Locations (1):
- Prentice Women's Hospital - Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: ACOG Solutions for the Surgical Preparation of the Vagina — https://www.ncbi.nlm.nih.gov/pubmed/23963423

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control (Povidone Iodine) | Intervention (4% Chlorhexidine Gluconate)
Started | 66 | 68
Completed | 63 | 60
Not Completed | 3 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control (Povidone Iodine) | Intervention (4% Chlorhexidine Gluconate) | Total
Number analyzed (Participants) | 63 | 60 | 123
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 59 | 59 | 118
  >=65 years | 4 | 1 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (10) | 44 (9) | 45 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 60 | 123
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 9 | 17
  White | 41 | 39 | 80
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 10 | 20
Region of Enrollment [Number; unit: participants]
  United States | 63 | 60 | 123

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Vaginal or Urinary Symptoms After Surgery, Assessed by Validated Questionnaire (Modified PRO-CTCAE)
Description: To determine and compare the number of participants with vaginal or urinary symptoms after treatment with chlorhexidine gluconate versus povidone iodine vaginal cleansing solutions.
Time Frame: Day of surgery to 24-48 hours after surgery
Population: Number of participants in control and active groups
Measure: Count of Participants; unit: Participants
Arm/Group | Control (Povidone Iodine) | Intervention (4% Chlorhexidine Gluconate)
Number analyzed (Participants) | 63 | 59
Participants
  Vaginal dryness | 4 | 11
  Vaginal burning | 8 | 25
  Unusual vaginal discharge | 10 | 14
  Pain of burning with urination | 9 | 17
  Vaginal itchiness | 7 | 7

ADVERSE EVENTS:
Time Frame: Data were collected for each patient immediately postoperatively to 24-48 hours postoperatively.
Description: The survey of vaginal & urinary symptoms used in this study was designed using the PRO-CTCAE (Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events) created by the NIH & NCI 7. The language & format of the PTO-CTCAE questions have been cognitively tested. Questions on vaginal burning and itching were investigator-developed items using similar language as the PRO-CTCAE, since these adverse events were not contained in the PRO-CTCAE item library.
Arm/Group | Control (Povidone Iodine) | Intervention (4% Chlorhexidine Gluconate)
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/60
Other Adverse Events (participants affected / at risk) | 0/63 | 1/59
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (Povidone Iodine) (N=63) | Intervention (4% Chlorhexidine Gluconate) (N=59)
Severe Swelling (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Genitourinary - One patient in the chlorhexidine group reported severe vulvar swelling that resolved within 24-48 hours after exposure

LIMITATIONS AND CAVEATS:
Single-blinded design. Present study included participants undergoing hysteroscopic procedures these procedures themselves may certainly influence postoperative irritative symptoms. Loss of follow-up both immediately and 24-48 hours postoperative.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-09): https://cdn.clinicaltrials.gov/large-docs/59/NCT03305159/Prot_SAP_000.pdf